CLINICAL TRIAL: NCT01046019
Title: Measurement of Early Bone Loss Around a Total Hip Arthroplasty. A Prospective Trial With Dual Energy X-ray Absorptiometry.
Brief Title: Measurement of Early Bone Loss Around a Total Hip Arthroplasty
Acronym: DXACorail
Status: Completed | Type: Observational
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Berte Bøe, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Other Study IDs: 35-07122b 1.2007.896
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2010-01

CONDITIONS: Coxarthrosis
Keywords: DXA; Hip; Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Research with DXA has shown the pattern of bone remodelling around an implant. The baseline and reference value for such calculations is the first measurement after the operation. The baseline measurement is performed at different time from study to study. If there is a rapid bone loss the first weeks after an operation, this will influence the reference value and then the results. To evaluate DXA as a method we decided to set up a study with 3 DXA measurements within the first 2 weeks. Our hypothesis is that there is a rapid bone loss the first 2 weeks after operation and that timing of the first post operative measurement will influence the later results.

DETAILED DESCRIPTION:
Dual x-ray absorptiometry (DXA) has become the most used and proven to be a precise method to investigate changes in bone mass density (BMD). Research with DXA has shown the pattern of bone remodelling around an implant. Results from implant studies are often presented as changes in BMD as a function of time. The baseline and reference value for such calculations is the first measurement after the operation. The most pronounced bone loss after implantation of hip prosthesis usually comes within 3 months. The baseline measurement is performed at different time from study to study. If there is a rapid bone loss the first weeks after an operation, this will influence the reference value and then the results. To evaluate DXA as a method we decided to set up a study with 3 DXA measurements within the first 2 weeks.

We included 23 patients operated with total hip prosthesis (THP). They were measured with DXA at 1, 5 and 14 days, 3 and 12 months after the operation. Results were given in percent (+/-SD) for each Gruen zone. There were no changes in bone density between the first 3 measurements. In all zones, except zone 1, the lowest BMD was measured after 3 months. We concluded that DXA measurements done within 14 days after the operation can be used as reference measurements for later follow ups.

ELIGIBILITY:
Inclusion Criteria:

* degenerative hip osteoarthritis

Exclusion Criteria:

* metastasis to bone
* dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with degenerative hip osteoarthritis decided for operation with total hip arthroplasty.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nordsletten, Professor, Study Director — Ullevaal University Hospital; Berte G Bøe, MD, Principal Investigator — Ullevaal University Hospital